CLINICAL TRIAL: NCT01579175
Title: The Effect of Gum Chewing on Postoperative Ileus After Gynecologic Surgery.
Acronym: GumGyn
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Catherine Sewell, Principal Investigator, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NA_00036423
Record Dates: First submitted 2012-04-13; First posted 2012-04-17 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Postoperative Ileus
MeSH Terms: interventions — Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard postoperative care (No Intervention)
- Chewing gum arm (Experimental): Sugar free (extra, spearment) chewing gum given to the patient to chew during waking hours every four hours for 15 minutes
  Interventions: Other: Chewing gum

INTERVENTIONS:
Other: Chewing gum — Sugar Free (Extra spearment) gum given to chew every 4 hours during waking hours for 15 minutes.
  Other Names: Extra spearment sugar free gum
  Arms: Chewing gum arm

SUMMARY:
The investigators are randomizing patients to receive chewing gum (Extra Sugar Free, Spearment) every 4 hours during waking hours for 15 minutes versus standard postoperative care. The investigators then have them fill out a survey in house and 1 week after their surgery that record time to first flatus, hunger, toleration of clear liquids and food and some information about pain, satisfaction, and quality of life. The investigators contact them via phone and email a maximum of three times in order to collect this information. 30 days postoperatively the investigators also contact them and perform a chart review for any postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Undergoing benign gynecologic surgery via an exploratory laparotomy
* Capable of giving consent

Exclusion Criteria:

* Oromaxillary or mental disturbances that would make chewing gum dangerous with regards to mastication or aspiration
* Intubated or unconscious when leaving the OR
* Bowel resection performed at the time of surgery
* Active bowel disease (IBD, appendicitis, etc)
* Gynecologic malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Time to flatus | 30 days

SECONDARY OUTCOMES:
Postoperative ileus | 30 days
  Nausea, vomiting, abdominal distention two episodes of 100cc of emesis
time to discharge | 30 days
time to toleration of diet | 30 days
patient satisfaction | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A Sewell, MD, MPH, Principal Investigator — Johns Hopkins University; Amelia M Jernigan, MD, Study Chair — Johns Hopkins University; Grace Chen, MD, Study Director — Johns Hopkins Bayview
Locations (2):
- United States (2):
  - Johns Hopkins Bayview, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland

REFERENCES:
- [Derived] Jernigan AM, Chen CC, Sewell C. A randomized trial of chewing gum to prevent postoperative ileus after laparotomy for benign gynecologic surgery. Int J Gynaecol Obstet. 2014 Dec;127(3):279-82. doi: 10.1016/j.ijgo.2014.06.008. Epub 2014 Jul 21. PMID 25147092